CLINICAL TRIAL: NCT02480075
Title: Therapeutic Evaluation to Research Clinical Objectives Linking Genotypic and Phenotypic Associations With Pain Management Outcomes
Brief Title: Observational Study Linking Genetic Variants With Clinical Outcomes in Pain Management
Acronym: TROJAN
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Proove Bioscience, Inc. (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: PB010
Record Dates: First submitted 2015-06-15; First posted 2015-06-24 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Pain; Chronic Pain
Keywords: Genetic Variation; Genetic Polymorphism; Polymorphism, Single Nucleotide; Genetic Association Studies
MeSH Terms: conditions — Pain; Chronic Pain | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic pain: Observational ; Adult patients seeking medical treatment that have been diagnosed with chronic pain.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational Study only

SUMMARY:
The purpose of this study is to (a) evaluate the treatment approaches and changes in treatment regimens utilized by clinicians when genetic testing is performed in the clinic; and (b) create a patient data registry to identify genetic factors that influence treatment outcomes in pain management.

DETAILED DESCRIPTION:
Clinicians who treat pain have noted that the response to opioids and other pain medications varies widely among patients. Differences in the degree of pain stimulation and pain sensitivity, weight and age differences, prior opioid use and tolerance, as well as the differences in bioavailability of various opioid formulations have been cited as causes for the wide variability in analgesia seen with opioids. However, a significant component of chronic pain may also be explained by genetic polymorphisms. Genetic information may explain the variability of responses and help predict more effective (or less dangerous) treatments and medication choices and doses. By identifying the genetic risks and the most effective analgesic for an individual patient, clinicians may be able to improve the efficacy of the pain treatments and medications and decrease the risk of iatrogenically-induced overdose, addiction, and death.

The purpose of this study is to evaluate how currently available genetic tests are being implemented in a pain management setting and whether this information results in benefits to patient care. Chronic pain patients receiving routine medical visits for their care will complete validated questionnaires to measure pain levels, disability indices, mental health, and quality of life measurements at each clinical visit. Physicians will document any changes made to treatment regimens, including adjustments to medications or non-pharmacological treatments and improvements in pain, functional ratings, or patient satisfaction. Concomitantly, this study will use the collected genetic and clinical data to create a data registry in order to examine novel correlations and associations between single nucleotide polymorphisms and longitudinal datasets.

The results of this study will elucidate potential predictive variables of chronic pain development and/or treatment that will assist in making better healthcare decisions in the selection of treatment modalities and dosing of medications for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.
* Currently experiencing a chronic pain problem, with symptoms that have occurred within the last 30 days.

Exclusion Criteria:

* Severe hepatic or renal disease
* Significant diminished mental capacity that is unable to understand the protocol, surveys and questionnaires; unable to read/write English or Spanish
* Recent febrile illness that precludes or delays participation by more than 1 month
* Pregnancy or lactation
* Participation in a clinical study that may interfere with participation in this study
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be adult patients seeking treatment at the Pain Clinic at the University of Southern California, Keck School of Medicine, in Los Angeles. Patients will have a chronic pain diagnosis and are receiving routine medical visits for their care. Treatment includes pharmacological, non-pharmacological treatment, interventional or infusion procedures, including ketamine infusion.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Pain Numeric Rating Scale (NRS) | Up to 2 years
Pain Scores on the CSS-17 | Up to 2 years
  The Chronic Regional Pain Syndrome (CRPS) Severity Score (CSS-17) is used for patients with CRPS.
Function/Disability assessment on the Oswestry Disability Index (ODI) | Up to 2 years
  The ODI is used for patients with back or neck pain.
Function/Disability assessment on the Headache Impact Test (HIT-6) | Up to 2 years
  The HIT-6 is used for patients with headaches or migraines.
Health-Related Quality of Life assessment on the SF-12v2 | Up to 2 years
  The Short Form 12 item-version 2 (SF-12v2) is a generic assessment of health-related quality of life.
Presence and Severity of Generalized Anxiety Disorder on the GAD-2/GAD-7 | Up to 2 years
  The GAD-2 short screening tool consists of the first two questions of the GAD-7 scale.
Presence and Severity of Depression on the PHQ-2/PHQ-9 | Up to 2 years
  The PHQ-2 is a short screening tool for the PHQ-9.
Number of Participants that Experience of Adverse Events | Up to 5 years
Type of Adverse Events Experienced by Participants | Up to 5 years
Severity of Adverse Events Experienced by Participants | Up to 5 years
Changes in type of treatments selected for participants | Up to 5 years
Changes in medication dosage for the participants | Up to 5 years
Changes in the frequency of urine drug screens | Up to 5 years

SECONDARY OUTCOMES:
The Session Rating Scale as a measure of the Patient-provider alliance | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Richeimer, M.D., Principal Investigator — University of Southern California
Locations (1):
- Pain Clinic at University of Southern California Keck Medical Center, Los Angeles, California, United States